CLINICAL TRIAL: NCT05589766
Title: N-DOSE: A Dose Optimization Trial of Nicotinamide Riboside in Parkinson's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Collaborators: University of Bergen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2022/426716
Record Dates: First submitted 2022-10-13; First posted 2022-10-21 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Parkinson Disease
Keywords: Parkinson's disease; NAD metabolism; Mitochondria; Nicotinamide Riboside
MeSH Terms: conditions — Parkinson Disease | interventions — nicotinamide-beta-riboside

STUDY DESIGN:
Intervention Model Description: Randomized double-blinded placebo-controlled study. 80 participants randomized in 1:1:2 ratio to either: 1. Placebo (n=20), 2. NR 1000mg for 3 months (n=20), 3. Dose escalation group: NR 1000mg 1st month, NR 2000mg 2nd month, NR 3000mg 3rd month (n=40).
Who Masked: Participant, Care Provider, Investigator
Masking Description: Both participants and all investigators are blinded during the trial and during data analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo, no active ingredients. Administered in tablet form twice daily for the duration of the trial (12 weeks).
  Interventions: Other: Placebo
- Dietary Supplement: NR 1000mg group (Experimental): Nicotinamide Riboside 1000mg total daily. Administered in capsule form in doses of 500mg twice daily for the duration of the trial (12 weeks).
  Interventions: Dietary Supplement: Nicotinamide Riboside
- Dietary Supplement: NR dose escalation group (Experimental): Nicotinamide Riboside dose escalation group: 1000mg NR daily in doses of 500mg twice daily (week 1 - week 4), 2000mg NR daily in doses of 1000mg twice daily (week 5 - week 8), 3000mg NR daily in doses of 1500mg twice daily (week 9 - week 12).
  Interventions: Dietary Supplement: Nicotinamide Riboside

INTERVENTIONS:
Dietary Supplement: Nicotinamide Riboside — Nicotinamide Riboside supplementation up to 3000mg daily in total.
  Other Names: Niagen; NR
  Arms: Dietary Supplement: NR 1000mg group; Dietary Supplement: NR dose escalation group
Other: Placebo — Placebo tablet identical in taste, form and appearance to NR tablets, administered twice daily for a total of 12 weeks.
  Arms: Placebo

SUMMARY:
N-DOSE is a double-blinded placebo-controlled randomized trial aiming to determine the optimal biological dose (OBD) of nicotinamide riboside (NR), in individuals with Parkinson's disease (PD).

The investigators recently reported the NADPARK study (ClinicalTrials.gov: NCT03816020), a phase I randomized, double-blinded trial, assessing the tolerability, cerebral bioavailability and molecular effects of NR therapy, 1000mg daily, in PD. The NADPARK study showed that NR 1000mg daily was well tolerated and led to a significant, but variable, increase in cerebral NAD (nicotinamide adenine dinucleotide) levels (measured by 31phosphorous magnetic resonance spectroscopy, 31P-MRS) and related metabolites in the cerebrospinal fluid (CSF). NR recipients showing increased brain NAD levels exhibited altered cerebral metabolism, measured by 18fluoro-deoxyglucose positron emission tomography (FDG-PET), and this was associated with mild clinical improvement. The results of the NADPARK trial nominate NR as a potential neuroprotective therapy for PD, warranting further investigation in larger trials. The investigators recently conducted the NR-SAFE safety trial comparing 3000mg NR to placebo in 20 participants with PD over 4 weeks (NCT: NCT05344404) which showed no moderate or severe adverse events, and no signs of acute toxicity.

Due to the variability in response to NR in the NADPARK trial, the N-DOSE study will investigate the response to escalating doses of NR from 1000 mg to 3000 mg over 12 weeks, in order to ascertain if NR dose escalation beyond 1000 mg per day is biologically meaningful in Parkinson's disease.

DETAILED DESCRIPTION:
N-DOSE is a double-blinded placebo-controlled randomized trial aiming to determine the optimal biological dose (OBD) of nicotinamide riboside (NR), in individuals with Parkinson's disease (PD).

Individuals with PD (n = 80) will be recruited starting November 2022. Participants will be randomized 1:1:2 to either placebo group (PL-group; n = 20) or NR 1000mg daily (DS-group; n = 20) for 12 weeks or to a dose-escalation group (DE-group) where NR 1000mg daily will be administered week 1-4, NR 2000mg daily week 5-8 and NR 3000mg daily week 9-12 (n =40). Both the participants and the investigators will be blinded.

- Primary Objective: To compare the effect of orally administered nicotinamide riboside (NR), escalated to 1500 mg twice per day (3000 mg/day) in the dose escalation group (DE-group) - versus stable dosing of 500 mg twice per day (1000 mg/day) in the dose-stable group (DS-group) on cerebral NAD levels, at week 12.

* Secondary Objectives:

  * To assess the dose-response relationship between NR dose (1000 mg, 2000 mg, 3000 mg per day) and changes in cerebral NAD levels from baseline to weeks 4, 8 and 12.
  * To compare the effectiveness of orally administered nicotinamide riboside (NR) 1500 mg twice per day versus 500 mg twice per day in augmenting the NAD-metabolome in the central nervous system (CNS) at week 12.
* Safety Objectives

  -- Determine the safety and tolerability of NR doses 2000 mg and 3000 mg daily in PD, measured by the frequency and severity of adverse events.
* Exploratory Objectives:

  * Neuroimaging

    * To compare the effect of orally administered NR in the DE-group versus DS-group on the NR related metabolic pattern (NRRP) expression at week 12.
    * To assess the dose-response relationship between NR dose (1000 mg, 2000 mg, 3000 mg per day) and changes in NRRP expression from baseline to weeks 4, 8 and 12.
    * To compare the effect of orally administered NR DE-group versus DS-group on the PD-related pattern (PDRP) expression at week 12.
    * To assess the dose-response relationship between NR dose (1000 mg, 2000 mg, 3000 mg per day) and changes in PDRP expression from baseline to weeks 4, 8 and 12.
  * Metabolism & molecular markers

    * To compare the effect of orally administered NR in the DE-group versus DS-group on the NAD metabolome* in the blood, urine and central nervous system (CNS) at week 12.
    * To assess the dose-response relationship between NR dose (1000 mg, 2000 mg, 3000 mg per day) and changes in the NAD metabolome* in blood and urine from baseline to weeks 4, 8 and 12.
    * To compare the effect of orally administered NR in the DE-group versus DS-group on serum and CSF inflammatory markers at week 12.
    * To assess the dose-response relationship between NR dose (1000 mg, 2000 mg, 3000 mg per day) and changes in serum inflammatory markers from baseline to weeks 4, 8 and 12.
  * Clinical - motor & non motor symptom severity, quality of life

    * To compare the effect of orally administered NR in the DE-group versus DS-group on clinical severity of PD symptoms at week 12.
    * To assess the dose-response relationship between NR dose (1000 mg, 2000 mg, 3000 mg per day) and change in clinical severity of PD symptoms from baseline to weeks 4, 8 and 12.
    * To compare the effect of orally administered NR in the DE-group versus DS-group on severity of non-motor symptoms of daily living in PD at week 12.
    * To assess the dose-response relationship between NR dose (1000 mg, 2000 mg, 3000 mg per day) and change in severity of non-motor symptoms of daily living in PD from baseline to weeks 4, 8 and 12.
    * To compare the effect of orally administered NR in the DE-group versus DS-group on severity of motor aspects of experiences of daily living in PD at week 12.
    * To assess the dose-response relationship between NR dose (1000 mg, 2000 mg, 3000 mg per day) and changes in severity of motor aspects of experiences of daily living in PD from baseline to weeks 4, 8 and 12.
    * To compare the effect of orally administered NR in the DE-group versus DS-group on severity of PD motor symptoms at week 12.
    * To assess the dose-response relationship between NR dose (1000 mg, 2000 mg, 3000 mg per day) and changes in severity of PD motor symptoms from baseline to weeks 4, 8 and 12.
    * To compare the effect of orally administered NR in the DE-group versus DS-group on severity PD motor complications at week 12.
    * To assess the dose-response relationship between NR dose (1000 mg, 2000 mg, 3000 mg per day) and changes in severity of PD motor complications from baseline to weeks 4, 8 and 12.
    * To compare the effect of orally administered NR in the DE-group versus DS-group on clinical severity of PD non-motor symptoms at week 12.
    * To assess the dose-response relationship between NR dose (1000 mg, 2000 mg, 3000 mg per day) and changes in clinical severity of PD non-motor symptoms from baseline to weeks 4, 8 and 12.
    * To compare the effect of orally administered NR in the DE-group versus DS-group on clinical severity of gastrointestinal non-motor dysfunction in PD at week 12.
    * To assess the dose-response relationship between NR dose (1000 mg, 2000 mg, 3000 mg per day) and changes in clinical severity of gastrointestinal non-motor dysfunction in PD from baseline to weeks 4, 8 and 12.
    * To compare the effect of orally administered NR in the DE-group versus DS-group on cognition at week 12.
    * To assess the dose-response relationship between NR dose (1000 mg, 2000 mg, 3000 mg per day) and changes in cognition from baseline to weeks 4, 8 and 12.
    * To compare the effect of orally administered NR in the DE-group versus DS-group on quality of life in PD at week 12.
    * To assess the dose-response relationship between NR dose (1000 mg, 2000 mg, 3000 mg per day) and changes in quality of life in PD from baseline to weeks 4, 8 and 12.
  * Hypothesis-generating or resource-dependent endpoints (may be reported in follow-up or secondary publications).

    * To compare the effect of orally administered NR in the DE-group versus DS-group on gene expression at week 12.
    * To assess the dose-response relationship between NR dose (1000 mg, 2000 mg, 3000 mg per day) and changes in gene expression from baseline to weeks 4, 8 and 12.
    * To compare the effect of orally administered NR in the DE-group versus DS-group on protein expression at week 12.
    * To assess the dose-response relationship between NR dose (1000 mg, 2000 mg, 3000 mg per day) and changes in protein expression from baseline to weeks 4, 8 and 12.
    * To compare the effect of orally administered NR in the DE-group versus DS-group on histone acetylation in PD at week 12.
    * To assess the dose-response relationship between NR dose (1000 mg, 2000 mg, 3000 mg per day) and changes in histone acetylation in PD from baseline to weeks 4, 8 and 12.
    * To compare the effect of orally administered NR in the DE-group versus DS-group on H3K27 and H4K16 histone acetylation in PD at week 12.
    * To assess the dose-response relationship between NR dose (1000 mg, 2000 mg, 3000 mg per day) and changes in on H3K27 and H4K16 histone acetylation in PD from baseline to weeks 4, 8 and 12.
    * To compare the effect of orally administered NR in the DE-group versus DS-group on the genomic distribution of H3K27 and H4K16 histone acetylation in PD at week 12.
    * To assess the dose-response relationship between NR dose (1000 mg, 2000 mg, 3000 mg per day) and changes in the genomic distribution of H3K27 and H4K16 histone acetylation in PD from baseline to weeks 4, 8 and 12.
    * To compare the effect of orally administered NR in the DE-group versus DS-group on folate and one-carbon metabolism in PD at week 12.
    * To assess the dose-response relationship between NR dose (1000 mg, 2000 mg, 3000 mg per day) and changes in folate and one-carbon metabolism in PD from baseline to weeks 4, 8 and 12.
    * To compare the effect of orally administered NR in the DE-group versus DS-group on methyl donors in PD at week 12.
    * To assess the dose-response relationship between NR dose (1000 mg, 2000 mg, 3000 mg per day) and changes in methyl-donors in PD from baseline to weeks 4, 8 and 12.
    * To compare the effect of orally administered NR in the DE-group versus DS-group on DNA methylation at week 12.
    * To assess the dose-response relationship between NR dose (1000 mg, 2000 mg, 3000 mg per day) and changes in methyl-donors in PD from baseline to weeks 4, 8 and 12.
    * To compare the effect of orally administered NR in the DE-group versus DS-group on synthesis of neurotransmitters in PD at week 12.
    * Determine whether NR-therapy affects the gut microbiome in a dose-responsive manner at week 12.
    * To compare the effect of orally administered NR in the DE-group versus DS-group on the gut metabolome at week 12.
    * To compare the effect of orally administered NR in the DE-group versus DS-group on the sense of smell at week 12.
    * To determine the safety and tolerability of NR at a dose of 1000 mg, 2000 mg, and 3000 mg per day in PD.
* Procedures:

All participants will attend study visits at Baseline, week 4, week 8 and week 12. The study visits will consist of the following:

* Assessment by one of the neurologists involved in the study including MDS-UPDRS
* Clinical testing with MDS-NMS, MoCA, EQ-5L and modified GIDS-PD by one of the study nurses involved in the sudy
* 31P-MRS, 1H-MRS and FDG-PET scan.
* Physical examination and measurement of vital signs
* Routine blood tests
* Urine sample collection
* Fecal sample collection
* Cerebrospinal fluid collection will be performed at Baseline and week 12

ELIGIBILITY:
Inclusion Criteria:

* Clinically established diagnosis of idiopathic PD according to the MDS criteria.
* 123I-Ioflupane dopamine transporter imaging (DAT-scan) confirming nigrostriatal degeneration.
* Hoehn and Yahr score < 4 at enrolment.
* Age ≥ 40 years at the time of enrollment.
* Able to undergo lumbar punction.
* Able to undergo MRI.

Exclusion Criteria:

* Dementia or other neurodegenerative disorder at baseline visit.
* Diagnosed with atypical parkinsonism (progressive supranuclear palsy (PSP), multiple system atrophy (MSA), corticobasal degeneration (CBD)) or vascular parkinsonism.
* Any psychiatric disorder that would interfere with compliance in the study.
* Metabolic, neoplastic, or other physically or mentally debilitating disorder at baseline visit.
* Use of high dose vitamin B3 supplementation within 30 days of enrollment.

Ages: 40 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2023-01-23 (Actual); Primary Completion 2025-04-22 (Actual); Study Completion 2025-04-22 (Actual)

PRIMARY OUTCOMES:
Cerebral NAD levels measured by 31P-MRS | 12 weeks for primary analysis. 4, 8 and 12 weeks for secondary analysis.
  Change in cerebral NAD/ATP-α ratio measured by 31 Phosphorus magnetic resonance spectroscopy (31P-MRS) in the posterior brain (encompassing the occipital, parietooccipital and posterior parts of the temporal cortex).

SECONDARY OUTCOMES:
CSF NAD or other metabolite of the NAD metabolome, measured by LC-MS | 12 weeks
  Change in the cerebrospinal fluid (CSF) levels of NAD or other metabolites of the NAD metabolome*, measured by LC-MS.

OTHER OUTCOMES:
Safety, measured by the frequency and severity of adverse events | 12 weeks
  Number and severity of adverse events from baseline to week 12 across treatment groups and NR dose levels.
Expression of the Nicotinamide Riboside Related Pattern (NRRP). | 12 weeks for primary analysis. 4, 8 and 12 weeks for secondary analysis.
  Change in NRRP expression, measured by FDG-PET.
Expression of the Parkinsons Disease Related Pattern (PDRP). | 12 weeks for primary analysis. 4, 8 and 12 weeks for secondary analysis.
  Change in PDRP expression, measured by FDG-PET.
NAD metabolites in blood, urine and CSF | 12 weeks
  Change in levels of NAD metabolites in blood, urine and CSF, measured by HPLC-MS and/or the NADMed method.
NAD metabolites in blood and urine | 4, 8 and 12 weeks
  Change in levels of NAD metabolites in blood and urine, measured by HPLC-MS and/or the NADMed method.
Inflammatory cytokines in serum and CSF | 12 weeks
  Change in inflammatory cytokines in serum and CSF, measured by ELISA.
Inflammatory cytokines in serum | 4, 8 and 12 weeks.
  Change in inflammatory cytokines in serum, measured by ELISA.
Total MDS-UPDRS score | 12 weeks for primary analysis. 4, 8 and 12 weeks for secondary analysis.
  Change in the total MDS-UPDRS score in the ON-medication state.
MDS-UPDRS part I score | 12 weeks for primary analysis. 4, 8 and 12 weeks for secondary analysis.
  Change in the MDS-UPDRS part I score in the ON-medication state.
MDS-UPDRS part II score | 12 weeks for primary analysis. 4, 8 and 12 weeks for secondary analysis.
  Change in the MDS-UPDRS part II score in the ON-medication state.
MDS-UPDRS part III score | 12 weeks for primary analysis. 4, 8 and 12 weeks for secondary analysis.
  Change in the MDS-UPDRS part III score in the ON-medication state.
MDS-UPDRS part IV score | 12 weeks for primary analysis. 4, 8 and 12 weeks for secondary analysis.
  Change in the MDS-UPDRS part IV score in the ON-medication state.
MDS-NMS score | 12 weeks for primary analysis. 4, 8 and 12 weeks for secondary analysis.
  Change in the total MDS-NMS score.
Modified GIDS-PD score | 12 weeks for primary analysis. 4, 8 and 12 weeks for secondary analysis.
  Change in the modified GIDS-PD score.
MoCA score | 12 weeks for primary analysis. 4, 8 and 12 weeks for secondary analysis.
  Change in the MoCA score.
EQ-5D-EL score | 12 weeks for primary analysis. 4, 8 and 12 weeks for secondary analysis.
  Change in the EQ-5D-5L score.
Gene expression, measured by RNA sequencing (RNAseq) | 12 weeks for primary analysis. 4, 8 and 12 weeks for secondary analysis.
  Change in gene expression, measured by RNA sequencing (RNAseq).
Protein expression, measured by LC-MS | 12 weeks for primary analysis. 4, 8 and 12 weeks for secondary analysis.
  Change in protein levels, measured by LC-MS.
Histone panacetylation, measured by immunoblotting | 12 weeks for primary analysis. 4, 8 and 12 weeks for secondary analysis.
  Change in histone panacetylation, measured by immunoblotting.
H3K27 and H4K16 histone acetylation | 12 weeks for primary analysis. 4, 8 and 12 weeks for secondary analysis.
  Changes in levels of H3K27 and H4K16 acetylation, measured by immunoblotting.
Genomic distribution of H3K27 and H4K16 histone acetylation | 12 weeks for primary analysis. 4, 8 and 12 weeks for secondary analysis.
  Change in the genomic distribution of H3K27 and H4K16 acetylation, measured by chromatin immunoprecipitation sequencing (ChIPseq).
Folate and one-carbon metabolism in blood and CSF | 12 weeks.
  Change in folate and one-carbon metabolites in blood and CSF, measured by HPLC-MS.
Folate and one carbon metabolism in blood | 4, 8 and 12 weeks.
  Change in folate and one-carbon metabolites in blood, measured by HPLC-MS.
Methyl-donors in blood and/or CSF | 12 weeks.
  Change in methyl-donors (e.g., SAM), measured by HPLC-MS, in the blood and/or CSF.
Methyl donors in blood | 4, 8 and 12 weeks.
  To assess the dose-response relationship between NR dose (1000 mg, 2000 mg, 3000 mg per day) and changes in methyl-donors in PD from baseline to weeks 4, 8 and 12. Change in methyl-donors (e.g., SAM), measured by HPLC-MS, in the blood.
DNA methylation | 12 weeks for primary analysis. 4, 8 and 12 weeks for secondary analysis.
  Change in level and genomic distribution of DNA methylation, measured by Illumina Infinium MethylationEpic kit.
Neurotransmitters in CSF | 12 weeks.
  Change in neurotransmitters in CSF, measured by HPLC-MS.
Gut microbiome composition | 12 weeks.
  Change in gut microbiome composition, measured by metagenomics in fecal samples.
Fecal metabolomics | 12 weeeks.
  Change in fecal metabolomics, measured by LC-MS in fecal samples.
Sense of smell | 12 weeks.
  Change in sense of smell, measured by B-SIT score.

CONTACTS AND LOCATIONS:
Overall Officials: Charalampos Tzoulis, PhD, Principal Investigator — Neuro-Sysmed, Haukeland University Hospital and University of Bergen
Locations (1):
- Haukeland University Hospital, Bergen, Vestland, Norway

DOCUMENTS (2):
  • Study Protocol (2025-06-05): https://cdn.clinicaltrials.gov/large-docs/66/NCT05589766/Prot_000.pdf
  • Statistical Analysis Plan (2025-06-16): https://cdn.clinicaltrials.gov/large-docs/66/NCT05589766/SAP_001.pdf